CLINICAL TRIAL: NCT02970344
Title: Improving Health Engagement and Lifestyle Management for Breast Cancer Survivors With Diabetes
Brief Title: I HEAL for Breast Cancer Survivors With Diabetes
Acronym: I HEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00073234
Record Dates: First submitted 2016-10-21; First posted 2016-11-22 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Diabetes
Keywords: Coping Skills Training; Diabetes Education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Coping Skills training (DCST) (Experimental): Twelve sessions are delivered over 6 months using a faded contact model involving 6 weekly sessions, 3 biweekly sessions and 3 monthly sessions.
  Interventions: Behavioral: Diabetes Coping Skills Training (DCST)
- Diabetes Education (No Intervention): one 60 minute diabetes education session.

INTERVENTIONS:
Behavioral: Diabetes Coping Skills Training (DCST) — Diabetes Coping Skills Training (DCST) consist of twelve 50 minutes sessions delivered over 6 months using a faded contact model ( 6 weekly session, 3 biweekly sessions and 3 monthly sessions)
  Arms: Diabetes Coping Skills training (DCST)

SUMMARY:
The proposed randomized clinical trial evaluates a diabetes coping skills training (DCST) intervention for improving breast cancer survivors' abilities to manage symptoms and adhere to recommended diabetes self-management. The telephone-based DCST protocol integrates three key strategies to reduce symptoms and improve diabetes self-management: coping skills training for managing symptoms, adherence skills training, and healthy lifestyle skills training. The investigator will test the effects of the DCST intervention by comparing it to diabetes education alone. Physical symptoms, psychological distress, diabetes self-management behaviors, and self-efficacy for managing symptoms and diabetes self-management will be assessed at baseline and 3, 6, and 12 months. Physical activity (i.e., daily steps and distance) will be assessed using wireless activity trackers and data will be obtained from home blood glucose monitoring devices. Glycosylated hemoglobin (HbA1c) will be assessed at baseline, 6, and 12 months.

DETAILED DESCRIPTION:
Together, breast cancer and type 2 diabetes represent a public health crisis. Approximately 20% of the 3.1 million breast cancer survivors in the U.S. have type 2 diabetes, and this number is expected to grow. Breast cancer survivors who have type 2 diabetes are at high risk for cancer recurrence, serious health complications, and premature death. Breast cancer survivors with type 2 diabetes experience more severe, disabling symptoms and psychological distress relative to breast cancer survivors without diabetes. For breast cancer survivors with type 2 diabetes, maintaining glycemic control is critical for decreasing symptoms and preventing serious health problems. Important diabetes self-management strategies include physical activity, dietary modifications, medication, and blood glucose monitoring. Many breast cancer survivors with type 2 diabetes have difficulty maintaining these behaviors and achieving glycemic control. Physical symptoms and psychological distress are often barriers to engaging in diabetes self-management. The proposed study evaluates a novel diabetes coping skills training (DCST) intervention for improving breast cancer survivors' abilities to manage symptoms and adhere to recommended diabetes self-management. The telephone-based DCST protocol is based on our prior work and integrates three key theory-based strategies: coping skills training for managing symptoms, adherence skills training, and healthy lifestyle skills training. The proposed randomized clinical trial (N=230) will test the effects of the DCST intervention by comparing it to diabetes education alone. Physical symptoms, psychological distress, diabetes self-management behaviors, and self-efficacy will be assessed at baseline and 3, 6, and 12 months. Physical activity will be assessed using wireless activity trackers and data will be obtained from home blood glucose monitoring devices. Glycosylated hemoglobin (HbA1c) will be assessed at baseline, 6, and 12 months. The proposed study addresses a critical gap in the care of breast cancer survivors by evaluating a novel behavioral intervention that aims to improve the management of symptoms, adherence, and glycemic control in breast cancer survivors with type 2 diabetes. The findings of this study could lead to significant improvements in clinical care and beneficial outcomes for breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Stage I to III breast cancer,
* diagnosis of diabetes mellitus type 2
* completed local definitive treatment (i.e., surgical treatment, chemotherapy and/or radiation therapy),
* physician verification of ability to participate in the intervention,
* English speaking.

Exclusion Criteria:

* <21 years of age,
* severe cognitive or hearing impairment,
* unable to provide meaningful consent (i.e., impairment such that descriptions of the research are not clearly understood),
* presence of a health problem that precludes safe participation in the intervention.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in physical symptoms | baseline, 3 months, 6 months and 12 months
  The Checklist measures the severity of different symptoms (e.g., pain, fatigue, numbness and tingling) associated with illness and disease.
Change in psychological distress | baseline, 3 months, 6 months and 12 months
  The eight-item Patient Reported Outcomes Information System (PROMIS).
Change in psychological distress | baseline, 3 months, 6 months and 12 months
  Anxiety will be assessed using the seven-item GAD-7 Scale.

SECONDARY OUTCOMES:
Accessing change in Diabetes self-management behaviors via self reported medication adherence | Baseline to 12 months
  Participants who receive DCST will exhibit greater improvements in medication adherence compare to the education group.
Accessing change in Diabetes self-management behavior via Barriers to taking medication | Baseline to 12 months
  Participants who receive DCST will exhibit greater improvements in medication adherence compare to the education group.
Accessing change in Diabetes self-management behavior via Adherence to diabetes self-management behaviors | Baseline to 12 months
  Participants who receive DCST will exhibit greater improvements in physical activity, dietary patterns, medication adherence, and adherence to blood glucose monitoring compare to the education group.
Accessing change in Diabetes self-management behavior via Use of home blood glucose monitoring | Baseline, 6 months and 12 months
  Participants who receive DCST will exhibit greater improvements in adherence to blood glucose monitoring compare to the education group.
Improved glycemic control | Baseline, 6 months and 12 months
  Participants who receive DCST will show greater improvements in HbA1c compared to the diabetes education alone.
Change in self-efficacy | Baseline, 6 months and 12 months
  This contains 5 items that inquire about patients' certainty about degree of pain control, pain during daily activities, controlling pain during sleep, and making pain reductions without extra medication.
Change in Physical Activity | Baseline, 6 months and 12 months
  Patient-reported physical activity will be assessed using the well-validated Community Healthy Activities Model Program for Seniors (CHAMPS).
  Participants who receive DCST will show improved self efficacy for managing symptoms and diabetes self-management compared to the diabetes education alone.
Assessing change in Physical Activity | Baseline, 6 months and 12 months
  Wireless activity tracking devices will be used to assess daily steps and distance.
  Participants who receive DCST will show improved self efficacy for managing symptoms and diabetes self-management compared to the diabetes education alone.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Shelby RA, Dorfman CS, Arthur SS, Bosworth HB, Corsino L, Sutton L, Owen L, Erkanli A, Keefe F, Corbett C, Kimmick G. Improving health engagement and lifestyle management for breast cancer survivors with diabetes. Contemp Clin Trials. 2020 May;92:105998. doi: 10.1016/j.cct.2020.105998. Epub 2020 Apr 11. PMID 32289471